CLINICAL TRIAL: NCT04160988
Title: A Single-center, Retrospective Study to Evaluate the Clinical Performance of Artificial Intelligence Medical Assisted Diagnostic Software (VeriSee DR) for Screening of Diabetic Retinopathy in Patients With Diabetes Mellitus
Status: Completed | Type: Observational
Sponsor: Acer Being Health Inc. (Industry)
Collaborators: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: QCR19002
Record Dates: First submitted 2019-11-07; First posted 2019-11-13 (Actual); Results first posted 2021-01-29 (Actual); Last update posted 2021-01-29 (Actual); Status verified 2021-01

CONDITIONS: Diabetic Retinopathy
MeSH Terms: conditions — Diabetic Retinopathy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study is to evaluate the clinical performance of VeriSee DR for DR screening from color fundus photography images in patients with diabetes mellitus. The sensitivity and specificity of VeriSee DR's automated image analysis for screening the diabetes retinopathy will be determined.

ELIGIBILITY:
Inclusion Criteria:

* Subjects enrolled in this study should meet all the following criteria.

  1. Subject with age ≥ 20 years old
  2. Subject with documented diagnosis of diabetes mellitus
  3. Subject with image taken by color fundus photography that meet the following requirement:

     * The resolution of image is 1024×1024 pixels or higher;
     * The angle view of image is 45 or 50 degree.
  4. Subject's image includes macula and optic nerve as judged by the ophthalmologist.

Exclusion Criteria:

* Subjects will be excluded if they meet any of the following criteria.

  1. The color fundus photography image previously used by VeriSee DR during the development process and pre-clinical test
  2. The macula, optic nerve, or other part in the image of color fundus photography is unclear to determine the disease condition as judged by the ophthalmologist.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Persons with diabetes, twenty years of age or older, who have been referred to an ophthalmologists for a dilated eye examination to detect diabetic retinopathy.
Sampling Method: Probability Sample
Enrollment: 703 (Actual)
Dates: Start 2019-12-16 (Actual); Primary Completion 2020-01-31 (Actual); Study Completion 2020-05-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

RESULTS

PARTICIPANT FLOW:
Groups:
- Test Group: A total of 703 subjects with at least one qualified color fundus photography image as determined by the ophthalmologist were enrolled in this study. All 703 subjects enrolled were included in the intended use population. A total of 703 qualified color fundus photography images from all enrolled subjects were included for effectiveness analysis. No subjects were excluded from the intended use population.
Period: Overall Study
Arm/Group | Test Group
Started | 703
Completed | 675
Not Completed | 28
Not completed — poor image quality | 28

BASELINE CHARACTERISTICS:
Groups:
- Intended Use Population: Intended Use Population
Arm/Group | Intended Use Population
Number analyzed (Participants) | 703
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.5 (13.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 354
  Male | 349
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Taiwan | 703

OUTCOME MEASURES:

1. Primary Outcome: Sensitivity
Description: To evaluate the clinical performance of VeriSee DR by determining the sensitivity.
  Sensitivity = 100% x TP/(TP+FN)
Time Frame: 2 months
Population: Of 703 subjects enrolled, VeriSee DR judged the images of 28 subjects (3.98%) as with insufficient image quality.
Measure: Number (95% Confidence Interval); unit: percent
Arm/Group | Intended Use Population
Number analyzed (Participants) | 675
percent | 95 [92.48 to 96.82]

2. Primary Outcome: Specificity
Description: To evaluate the clinical performance of VeriSee DR by determining the specificity.
  Specificity = 100% x TN/(TN+FP)
Time Frame: 2 months
Population: Of 703 subjects enrolled, VeriSee DR judged the images of 28 subjects (3.98%) as with insufficient image quality.
Measure: Number (95% Confidence Interval); unit: percent
Arm/Group | Test Group
Number analyzed (Participants) | 675
percent | 89.9 [85.37 to 96.43]

3. Secondary Outcome: Positive Predictive Values (PPV)
Description: To evaluate the clinical performance of VeriSee DR by determining the positive predictive values (PPV).
  Positive predictive value (PPV) =100% x TP/(TP+FP)
Time Frame: 2 months
Population: Of 703 subjects enrolled, VeriSee DR judged the images of 28 subjects (3.98%) as with insufficient image quality.
Measure: Number (95% Confidence Interval); unit: percent
Arm/Group | Test Group
Number analyzed (Participants) | 675
percent | 94.5 [91.97 to 96.47]

4. Secondary Outcome: Negative Predictive Values (NPV)
Description: To evaluate the clinical performance of VeriSee DR by determining the negative predictive values (NPV).
  Negative predictive value (NPV) = 100% x TN/(FN+TN)
Time Frame: 2 months
Population: Of 703 subjects enrolled, VeriSee DR judged the images of 28 subjects (3.98%) as with insufficient image quality.
Measure: Number (95% Confidence Interval); unit: percent
Arm/Group | Intended Use Population
Number analyzed (Participants) | 675
percent | 90.7 [86.23 to 94.07]

5. Secondary Outcome: Percentage of Participant Images With Insufficient Quality as Judged by VeriSee DR
Description: To determine the percentage of subjects' images with insufficient quality as judged by VeriSee DR.
  The percentage of subjects who have the images with insufficient quality as determined by VeriSee DR will be presented.
Time Frame: 2 months
Measure: Count of Participants; unit: Participants
Arm/Group | Intended Use Population
Number analyzed (Participants) | 703
Participants | 28

ADVERSE EVENTS:
Time Frame: this study is a retrospective study so there is no need to collect adverse event data.
Description: this study is a retrospective study so there is no need to collect adverse event data.
Arm/Group | Test Group
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2019-07-30): https://cdn.clinicaltrials.gov/large-docs/88/NCT04160988/Prot_000.pdf